CLINICAL TRIAL: NCT04631640
Title: Prognostic Model of HCV-related Disease Progression After DAAs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Huixin, Assistant professor, Peking University People's Hospital
Other Study IDs: PHSC-1
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: HCV
Keywords: HCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — 5 ml blood sample would taken at each follow-up, and used to test ALT, AST, ALP, AFP and HCV RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigator would conduct an ambispective cohort study to build a prediction model of HCV-related disease after DAAs.

DETAILED DESCRIPTION:
The emergence of direct antiviral agents (DAAs) makes it possible to cure HCV, and the sustained virological response (SVR) rate is up to 90% after DAAs therapy. However, the acquisition of SVR does not mean the cure of HCV-related diseases, some patients still developed liver cirrhosis, liver cancer and other diseases after achived SVR by DAAs therapy.In this study the investigator would like to bulid a prediction model of HCV-related disease after DAAs by conducting an ambispective cohort study. The participants of this study would be adult patients (≥18 years old) with chronic HCV infection and have received DAA therapy, the investigator would retrospectively collected DAA therapy-related information, and follow-up all the enrolled participants every 6 months to observe their liver-related disease outcomes (composite liver outcome, including liver-related deaths, hepatocellular carcinoma, liver decompensation, and liver transplantation).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years old) with chronic HCV infection that were HCV RNA positive;
* have received DAA treatment;
* would like to adhere to the follow-up

Exclusion Criteria:

* lack of HCV treatment information;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with chronic HCV infection that were HCV RNA positive and have received DAA therapy were included, former hcv treatment information and sustained virologic response data were collected restropectively, liver-related events including liver-related deaths, HCC, liver decompensation, and liver transplantation were collected restropectively and prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of composit liver-related events | through study completion, an average of 2 year
  Composite liver outcomes, including liver-related deaths, hepatocellular carcinoma, liver decompensation, or liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Huixin Liu, Ph.D., Principal Investigator — Peking University People's Hospital